CLINICAL TRIAL: NCT05493683
Title: A Single Arm, Open Label, Multiple Center, Prospective Study of Disitamab Vedotin Combined With Tislelizumab in HER2 Positive Advanced Colorectal Cancer Failed at Least Two Lines of Systemic Treatment.
Brief Title: Disitamab Vedotin Combined With Tislelizumab in Advanced HER2 Positive Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-G 07
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Cancer; Antibody Drug Conjugate; Disitamab Vedotin; Tislelizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — disitamab vedotin; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of Disitamab Vedotin and Tislelizumab (Experimental): Disitamab Vedotin 2.0mg/kg q2w+Tislelizumab 400mg q6w. The treatment of Disitamab Vedotin + Tislelizumab will continue until the tumor progression confirmed by imaging, or up to 2 years, or intolerable toxic reactions, or other conditions determined by the researchers.
  Interventions: Drug: Disitamab vedotin; Drug: Tislelizumab

INTERVENTIONS:
Drug: Disitamab vedotin — 2.0mg/kg，q2w
  Other Names: RC48
Drug: Tislelizumab — 400mg，q6w

SUMMARY:
Among patients with colonrectal cancer, 5% were HER-2 positive, but the immunohistochemical results were mostly HER-2 2 +, which did not meet the indications of HER-2 targeting drugs. Disitamab Vedotin , which was listed in China last year, achieved similar results in HER-2 2+ and 3+, according to a clinical trial for breast cancer, suggesting that patients with colonrectal cancer may benefit from it. Tislelizumab is a PD-1 monoclonal antibody, which has been approved for a variety of tumors. It was reported that anti-HER-2 treatment can improve the tumor immune microenvironment and improve the efficacy of immunotherapy. At the same time, our previous studies showed that anti-PD-1 combined with Disitamab Vedotin can significantly inhibit the growth of colon tumor in mice. Therefore, Disitamab Vedotin and Tislelizumab were used in this study. This prospective clinical trial may bring new hope for the treatment of HER-2 positive CRC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the consents voluntarily;
2. All genders, age 18 or above;
3. Histological or cytological documentation of local advanced or metastatic unresectable colorectal carcinoma;
4. Patients with HER-2 overexpression (HER-2 IHC 2+ or IHC 3+) detected by immunohistochemistry; Resampling is recommended for samples over 3 years.
5. Subjects must have failed at treatments including fluoropyrimidine, oxaliplatin and irinotecan; For adjuvant or neoadjuvant chemotherapy, if disease progression occurs during treatment or within 6 months after treatment, it will be recorded as a first-line treatment;
6. Patients who have used anti-PD-1 or anti-PD-L1 inhibitors can be selected after stopping the treatment for more than 6 months; Patients who have used other anti HER-2 drugs with different mechanisms can be selected.
7. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.is necessary
8. Life expectancy of at least 3 months.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
10. Have sufficient heart, lung, liver and kidney functions, and the laboratory examination within 14 days before screening meets the following indicators:

    i. Hemoglobin Hb ≥ 90 g/L ii. Neutrophil count ANC ≥ 1.5*10^9 /L iii. Platelet count PLT ≥ 80*10^9 /L iv. Albumin ALB ≥ 35 g/L v. Alanine aminotransferase ALT and aspartate aminotransferase AST ≤ 2.5 times the upper limit of the normal range, and liver metastasis patients ≤ 5 times the upper limit of the normal range.

    vi. Total bilirubin ≤ 1.5 times, or 2 times the upper limit of normal. vii. Creatinine Scr ≤ upper limit of normal range. viii. Prothrombin: PT-INR ≤ 2.3 or PT < 6 seconds compared with normal control
11. Subjects must complete the treatment and follow-up on schedule. according to the research plan.
12. No brain metastasis, no spinal cord compression.
13. Subjects agree to use blood samples for study analysis.
14. Women of childbearing age must be negative in pregnancy test and willing to take effective contraceptive measures during the study period.

Exclusion Criteria:

1. Subjects are severe malnutrition or need tube feeding.
2. Major surgery has been performed within 30 days before treatment.
3. Previous treatment with anti-PD-1 / PD-L1 inhibitor, anti-CTLA-4 inhibitor, ADC drugs targeting HER-2 such as RC48 and T-DM1 within 6 months.
4. Other malignant tumors within 2 years and without cure (Except for patients with other early-stage tumors, after radical treatment, whom the researchers assess the recurrence risk of in the short term is small);
5. Subjects have active autoimmune system diseases that need systemic hormone therapy or anti autoimmune drug therapy.
6. Subjects with immunodeficiency or receiving systemic steroid therapy (prednisone > 10 mg / day or other equivalent drugs) or other forms of immunosuppressive therapy 7 days before the first dose of combination therapy in this study;
7. Subjects with active infection and still need systemic treatment 7 days before the first dose of therapy in this study.
8. Subjects with uncontrollable systemic diabetes.
9. Subjects with interstitial lung disease, non infectious pneumonia or pulmonary fibrosis;
10. Subjects who have received allogeneic organ or stem cell transplantation in the past.
11. Subjects allergic to the drugs or related components involved in this study.
12. Participating in other interventional clinical studies.
13. The previous anti-tumor related adverses do not return to grade 1 in CTCAE before the first combination therapy.
14. Subjects who have uncontrolled hypertension by drugs, that is, systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg.
15. Thrombotic or hemorrhagic tendency or history within 60 days before the first medication, regardless of the severity.
16. Any serious or unstable medical condition#mental illness or known active alcohol or drug abuse or dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | up to 2 years
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR)

SECONDARY OUTCOMES:
Progression-free Survival(PFS) | From date of subjects until the date of first documented progression or death from any cause, whichever came first, assessed up to 24 months
  PFS was defined as the time from assignment to disease progression radiological/clinical or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.
Overall Survival (OS) | From assignment of the first subject until 32 death events observed, up to 2 years.
  OS is defined as the time from date of assignment to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Disease control rate (DCR) | up to 2 years
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD).
Safety and Feasibility | up to 2 years
  Safety is defined as the incidence of Grade 3-4 Treatment-Related Adverse Events (TRAEs) from the day of neoadjuvant therapy to 30 days after surgery or within 90 days after last neoadjuvant treatment. Feasibility of surgery is defined as the incidence of TRAEs causing surgery delay of ≥30 days and/or inoperable patients.Feasibility of surgery is defined as the incidence of TRAEs causing surgery delay of ≥30 days and/or inoperable patients.
Duration of Response (DOR) | up to 2 years
  DOR is defined as the time from randomization to disease progression or death in patients who achieve complete or partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Gu Yanhong, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (6):
- China (6):
  - Changzhou NO.2 People's Hospital, Changzhou, Jiangsu
  - The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, Huai'an, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - the Third Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Diagnosis And Treatment Guidelines For Colorectal Cancer Working Group CSOCOC. Chinese Society of Clinical Oncology (CSCO) diagnosis and treatment guidelines for colorectal cancer 2018 (English version). Chin J Cancer Res. 2019 Feb;31(1):117-134. doi: 10.21147/j.issn.1000-9604.2019.01.07. No abstract available. PMID 30996570
- [Background] Messersmith WA. NCCN Guidelines Updates: Management of Metastatic Colorectal Cancer. J Natl Compr Canc Netw. 2019 May 1;17(5.5):599-601. doi: 10.6004/jnccn.2019.5014. PMID 31117039
- [Background] Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, Aranda Aguilar E, Bardelli A, Benson A, Bodoky G, Ciardiello F, D'Hoore A, Diaz-Rubio E, Douillard JY, Ducreux M, Falcone A, Grothey A, Gruenberger T, Haustermans K, Heinemann V, Hoff P, Kohne CH, Labianca R, Laurent-Puig P, Ma B, Maughan T, Muro K, Normanno N, Osterlund P, Oyen WJ, Papamichael D, Pentheroudakis G, Pfeiffer P, Price TJ, Punt C, Ricke J, Roth A, Salazar R, Scheithauer W, Schmoll HJ, Tabernero J, Taieb J, Tejpar S, Wasan H, Yoshino T, Zaanan A, Arnold D. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016 Aug;27(8):1386-422. doi: 10.1093/annonc/mdw235. Epub 2016 Jul 5. PMID 27380959
- [Background] Piawah S, Venook AP. Targeted therapy for colorectal cancer metastases: A review of current methods of molecularly targeted therapy and the use of tumor biomarkers in the treatment of metastatic colorectal cancer. Cancer. 2019 Dec 1;125(23):4139-4147. doi: 10.1002/cncr.32163. Epub 2019 Aug 21. PMID 31433498
- [Background] Shirley M. Fruquintinib: First Global Approval. Drugs. 2018 Nov;78(16):1757-1761. doi: 10.1007/s40265-018-0998-z. PMID 30357594
- [Background] Oh DY, Bang YJ. HER2-targeted therapies - a role beyond breast cancer. Nat Rev Clin Oncol. 2020 Jan;17(1):33-48. doi: 10.1038/s41571-019-0268-3. Epub 2019 Sep 23. PMID 31548601
- [Background] Rakha EA, Pinder SE, Bartlett JM, Ibrahim M, Starczynski J, Carder PJ, Provenzano E, Hanby A, Hales S, Lee AH, Ellis IO; National Coordinating Committee for Breast Pathology. Updated UK Recommendations for HER2 assessment in breast cancer. J Clin Pathol. 2015 Feb;68(2):93-9. doi: 10.1136/jclinpath-2014-202571. Epub 2014 Dec 8. PMID 25488926
- [Background] Ruschoff J, Hanna W, Bilous M, Hofmann M, Osamura RY, Penault-Llorca F, van de Vijver M, Viale G. HER2 testing in gastric cancer: a practical approach. Mod Pathol. 2012 May;25(5):637-50. doi: 10.1038/modpathol.2011.198. Epub 2012 Jan 6. PMID 22222640
- [Background] Mar N, Vredenburgh JJ, Wasser JS. Targeting HER2 in the treatment of non-small cell lung cancer. Lung Cancer. 2015 Mar;87(3):220-5. doi: 10.1016/j.lungcan.2014.12.018. Epub 2015 Jan 8. PMID 25601485
- [Background] Siena S, Sartore-Bianchi A, Marsoni S, Hurwitz HI, McCall SJ, Penault-Llorca F, Srock S, Bardelli A, Trusolino L. Targeting the human epidermal growth factor receptor 2 (HER2) oncogene in colorectal cancer. Ann Oncol. 2018 May 1;29(5):1108-1119. doi: 10.1093/annonc/mdy100. PMID 29659677
- [Background] Valtorta E, Martino C, Sartore-Bianchi A, Penaullt-Llorca F, Viale G, Risio M, Rugge M, Grigioni W, Bencardino K, Lonardi S, Zagonel V, Leone F, Noe J, Ciardiello F, Pinto C, Labianca R, Mosconi S, Graiff C, Aprile G, Frau B, Garufi C, Loupakis F, Racca P, Tonini G, Lauricella C, Veronese S, Truini M, Siena S, Marsoni S, Gambacorta M. Assessment of a HER2 scoring system for colorectal cancer: results from a validation study. Mod Pathol. 2015 Nov;28(11):1481-91. doi: 10.1038/modpathol.2015.98. Epub 2015 Oct 9. PMID 26449765
- [Background] Sartore-Bianchi A, Trusolino L, Martino C, Bencardino K, Lonardi S, Bergamo F, Zagonel V, Leone F, Depetris I, Martinelli E, Troiani T, Ciardiello F, Racca P, Bertotti A, Siravegna G, Torri V, Amatu A, Ghezzi S, Marrapese G, Palmeri L, Valtorta E, Cassingena A, Lauricella C, Vanzulli A, Regge D, Veronese S, Comoglio PM, Bardelli A, Marsoni S, Siena S. Dual-targeted therapy with trastuzumab and lapatinib in treatment-refractory, KRAS codon 12/13 wild-type, HER2-positive metastatic colorectal cancer (HERACLES): a proof-of-concept, multicentre, open-label, phase 2 trial. Lancet Oncol. 2016 Jun;17(6):738-746. doi: 10.1016/S1470-2045(16)00150-9. Epub 2016 Apr 20. PMID 27108243
- [Background] Meric-Bernstam F, Hurwitz H, Raghav KPS, McWilliams RR, Fakih M, VanderWalde A, Swanton C, Kurzrock R, Burris H, Sweeney C, Bose R, Spigel DR, Beattie MS, Blotner S, Stone A, Schulze K, Cuchelkar V, Hainsworth J. Pertuzumab plus trastuzumab for HER2-amplified metastatic colorectal cancer (MyPathway): an updated report from a multicentre, open-label, phase 2a, multiple basket study. Lancet Oncol. 2019 Apr;20(4):518-530. doi: 10.1016/S1470-2045(18)30904-5. Epub 2019 Mar 8. PMID 30857956
- [Background] Sartore-Bianchi A, Lonardi S, Martino C, Fenocchio E, Tosi F, Ghezzi S, Leone F, Bergamo F, Zagonel V, Ciardiello F, Ardizzoni A, Amatu A, Bencardino K, Valtorta E, Grassi E, Torri V, Bonoldi E, Sapino A, Vanzulli A, Regge D, Cappello G, Bardelli A, Trusolino L, Marsoni S, Siena S. Pertuzumab and trastuzumab emtansine in patients with HER2-amplified metastatic colorectal cancer: the phase II HERACLES-B trial. ESMO Open. 2020 Sep;5(5):e000911. doi: 10.1136/esmoopen-2020-000911. PMID 32988996
- [Background] Nakamura Y, et al. TRIUMPH: Primary efficacy of a phase II trial of trastuzumab (T) and pertuzumab (P) in patients (pts) with metastatic colorectal cancer (mCRC) with HER2 (ERBB2) amplification (amp) in tumor tissue or circulating tumor DNA (ctDNA): a GOZILA sub-study. Annals of Oncology (2019) 30 (suppl_5): v198-v252.
- [Background] Strickler JH, et al. Trastuzumab and tucatinib for the treatment of HER2 amplified metastatic colorectal cancer (mCRC): Initial results from the MOUNTAINEER trial. Annals of Oncology (2019) 30 (suppl_5): v198-v252.
- [Background] Siena S, Di Bartolomeo M, Raghav K, Masuishi T, Loupakis F, Kawakami H, Yamaguchi K, Nishina T, Fakih M, Elez E, Rodriguez J, Ciardiello F, Komatsu Y, Esaki T, Chung K, Wainberg Z, Sartore-Bianchi A, Saxena K, Yamamoto E, Bako E, Okuda Y, Shahidi J, Grothey A, Yoshino T; DESTINY-CRC01 investigators. Trastuzumab deruxtecan (DS-8201) in patients with HER2-expressing metastatic colorectal cancer (DESTINY-CRC01): a multicentre, open-label, phase 2 trial. Lancet Oncol. 2021 Jun;22(6):779-789. doi: 10.1016/S1470-2045(21)00086-3. Epub 2021 May 4. PMID 33961795
- [Background] Sheng X, Yan X, Wang L, Shi Y, Yao X, Luo H, Shi B, Liu J, He Z, Yu G, Ying J, Han W, Hu C, Ling Y, Chi Z, Cui C, Si L, Fang J, Zhou A, Guo J. Open-label, Multicenter, Phase II Study of RC48-ADC, a HER2-Targeting Antibody-Drug Conjugate, in Patients with Locally Advanced or Metastatic Urothelial Carcinoma. Clin Cancer Res. 2021 Jan 1;27(1):43-51. doi: 10.1158/1078-0432.CCR-20-2488. Epub 2020 Oct 27. PMID 33109737
- [Background] Sheng XN, He ZS, Han WQ, et al. An Open-label, Single-arm, Multicenter, Phase Ⅱ Study of RC48 to Evaluate the Efficacy and Safety of Subjects With HER2 Overexpressing Locally Advanced or Metastatic Urothelial Cancer (RC48-C009) [EB/OL]. ASCO 2021, abstract 4584.
- [Background] Zhou L, Xu HY, Yan XQ, et al. Preliminary results of RC48 combined with toripalimab in patients with locally advanced or metastatic urothelial carcinoma RC48-C014[EB/OL]. ASCO 2021, abstract 4534.